CLINICAL TRIAL: NCT03965299
Title: Transcutaneous Tibial Nerve Stimulation in Patients With Acute Spinal Cord Injury to Prevent Neurogenic Detrusor Overactivity: A Nationwide Randomised, Sham-controlled, Double-blind Clinical Trial
Brief Title: Transcutaneous Tibial Nerve Stimulation in Acute Spinal Cord Injury
Acronym: TASCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other); Clinique Romande de Readaptation (Network); Rehab Basel (Other); Swiss Paraplegic Research, Nottwil (Network); BioMedical Research Forschungslabor für Urologie, University of Bern (Unknown); Translational Neuro-Urology Department of Biomedicine, University of Porto (Unknown); Center for Lower Urinary Tract Research School of Medicine, University of Pittsburgh (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019-00074
Record Dates: First submitted 2019-03-26; First posted 2019-05-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injury, Acute
Keywords: randomized, sham-controlled, double-blind trial; transcutaneous tibial nerve stimulation; spinal cord injury; neurogenic detrusor overactivity; neuromodulation; electrical stimulation; paraplegia; tetraplegia; urodynamics
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Quadriplegia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The only unmasked person involved in the trial is the operator who will be responsible for the daily application of the study intervention at the patient. The role of an operator can be occupied by a research assistant/study nurse or investigator not involved in the clinical management and assessment of clinical outcomes. Thus, patients and care providers involved with clinical assessments are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VERUM transcutaneous tibial nerve stimulation (TTNS) (Experimental)
  Interventions: Device: VERUM TTNS
- SHAM transcutaneous tibial nerve stimulation (TTNS) (Sham Comparator)
  Interventions: Device: SHAM TTNS

INTERVENTIONS:
Device: VERUM TTNS — * Daily 30-minute TTNS intervention is performed 5 days a week during a treatment period of 6-9 weeks, until 3-month post assessments
  * During a preparation phase of several minutes, sensory and motor thresholds are assessed and stimulation intensities are adjusted for the following 30-minute treatment phase
  Arms: VERUM transcutaneous tibial nerve stimulation (TTNS)
Device: SHAM TTNS — * Daily 30-minute SHAM intervention is performed 5 days a week during a treatment period of 6-9 weeks, until 3-month post assessments
  * During a preparation phase of several minutes, sensory and motor thresholds are assessed and stimulation intensities are adjusted for the following 30-minute treatment phase
  Arms: SHAM transcutaneous tibial nerve stimulation (TTNS)

SUMMARY:
Most patients with spinal cord injury (SCI) develop neurogenic lower urinary tract dysfunction (NLUTD), one of the most devastating sequelae of SCI which ultimately can lead to renal failure. We urgently need an intervention that prevents NLUTD before irreversible damage occurs. Neuromodulation procedures are a promising avenue so that we investigate the effect of transcutaneous tibial nerve stimulation (TTNS) in patients with acute SCI.

This nationwide randomized, sham-controlled, double-blind multicentre clinical trial includes all SCI centres in Switzerland (Basel, Nottwil, Sion, Zürich). Patients are randomly assigned to VERUM TTNS (active stimulation, n=57) and SHAM stimulation (n=57) groups in a 1:1 allocation using computer-generated permuted block randomisation lists stratified on study centre and lower extremity motor score. Daily 30-minute sessions are performed five times a week during an intervention period of 6-9 weeks. The primary outcome of this study is the success of TTNS to prevent neurogenic DO jeopardizing the upper urinary tract, assessed by urodynamics at 1 year after SCI or any earlier time point if DO treatment is necessary (study end). Secondary outcome measures are bladder diary parameters, clinical symptom scores assessed by standardized and validated questionnaires. Furthermore, neurophysiological and neuroimaging outcome measures are assessed as well as, biochemical and molecular changes. Tertiary outcome measure is the safety of TTNS.

Before the actual start of the TASCI RCT, start-up activities will include a piloting phase on groups of healthy volunteers and patients. The goal during this phase is to evaluate the feasibility of the experimental setup, in particular for the TTNS and SHAM intervention, but also to test the setup of the different pre and post assessments (e.g. neurophysiology and neuroimaging tests). Groups of up to 15 participants each will be enrolled in a few consecutive pilot studies allowing for fine tuning and small adaptations in between, if appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients with acute SCI (traumatic SCI and sudden onset (<7 days) non-traumatic SCI) within 40 days after injury
* Patients with acute SCI at cervical or thoracic level
* Willing to take part and follow the requirements of the TASCI protocol (up to one year after SCI)

  * no percutaneous tibial nerve stimulation (PTNS)
  * no functional electrical stimulation (FES), apart from upper limb FES
  * no electrical muscle stimulation (EMS)
* Informed Consent

Exclusion Criteria:

* Contraindications to the investigational product
* DO with contractions greater than 40 cmH2O at a bladder filling volume of less than 500mL at baseline visit
* Treatment with antimuscarinics or with mirabegron
* Known or suspected non-adherence, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another study with investigational drug or product within the 30 days preceding and during the present study
* Neuromodulation treatment for urological or bowel indication in the last six months or ongoing
* Botulinum toxin injections in the detrusor and/or urethral sphincter in the last six months
* Bilaterally absent tibial nerve compound muscle action potential (cMAP, amplitude < 1mV)
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Individuals especially in need of protection (according to Research with Human Subjects published by the Swiss Academy of Medical Sciences [www.samw.ch/en/News/News.html])
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Pre-existing or concomitant medical condition apart from SCI that might pose a safety issue or would interfere with interpretation of study results or study conduct (e.g. Parkinson's disease, neurodegenerative disorders including multiple sclerosis and amyotrophic lateral sclerosis, urological malignancies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The occurrence of neurogenic DO jeopardizing the upper urinary tract | up to 12 months after SCI
  Defined as composite measure: Urodynamic assessment establishing DO amplitude ≥40 cmH2O; or else initiation of DO treatment (with antimuscarinics and/or intradetrusor onabotulinumtoxinA injections)

SECONDARY OUTCOMES:
Volumetric changes during urodynamics and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  Cystometric capacity [mL], volume at first DO [mL], voided volume [mL] and post void residual [mL] as assessed by urodynamic measurement
Changes in bladder compliance [mL/cmH2O] during urodynamics and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
Pressure changes during urodynamics and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  Maximum DO amplitude [cmH2O], detrusor leak-point pressure [cmH2O], maximum detrusor pressure [cmH2O] during storage phase, maximum detrusor pressure [cmH2O] during voiding phase, detrusor pressure at maximum flow rate [cmH2O] as assessed by urodynamic measurement
Changes in maximum flow rate [mL/s] as assessed by urodynamics and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
Changes in vesicoureterorenal reflux (VUR) as assessed by videography during urodynamics and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
Changes in pelvic floor activity as assessed by electromyography (EMG) during urodynamics and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
Changes in bladder storage and voiding parameters and their relation to clinical outcomes | Baseline; once every 2 weeks during the TTNS intervention period; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  Assessed by a bladder diary
Changes in bowel diary parameters and their relation to clinical outcomes | Baseline; once every 2 weeks during the TTNS intervention period; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  Assessed by a bowel diary
Changes in International Prostate Symptom (IPSS) questionnaire and their relation to clinical outcomes | Baseline; once per week during the TTNS intervention period; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  The IPSS ("International Prostate Symptom Questionnaire") score is based on questions concerning urinary symptoms and quality of life (QoL). It consists of 8 items covering 7 urinary symptoms related dimensions (subscales) and 1 additional item assessing quality of life. Each item is rated on a 6-point scale (0=not at all; 5=almost always). The lowest possible score in the total IPSS score is 0 (asymptomatic); the highest possible score is 35 (symptomatic). The QoL index is rated on a 7-point scale, with 0 indicating "delighted" and 6 "terrible."
Changes in urinary symptoms as assessed by the Urinary Symptom Profile (USP) questionnaire and their relation to clinical outcomes | Baseline; once per week during the TTNS intervention period; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  The USP ("Urinary Symptom Profile") score is based on questions concerning urinary symptoms and their severity in males and females. It consists of 13 items covering 3 dimensions (subscales) with 7 overactive bladder (OAB), 3 stress urinary incontinence (SUI), and 3 low stream (LS) related items. Each item is rated on a 4-point scale. The lowest score is 0 (asymptomatic); the highest score is 3 (symptomatic).
Changes in Qualiveen questionnaire scores and their relation to clinical outcomes | Baseline; once per week during the TTNS intervention period; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  Qualiveen-30 assesses the Specific Impact of Urinary Problems (SIUP) on Quality of Life. It consists of 30 items covering 4 domains, namely inconvenience (9 questions), restrictions (8 questions), fears (8 questions), and impact on daily life (5 questions). Each item is rated on a 5-point ordinal scale (0=asymptomatic; 4=symptomatic). The index of the SIUP on Quality of Life is the mean of the four individual scores. The lowest possible overall score in the Qualiveen-30 is 0 (Urinary problems have no specific impact on QoL); the highest possible score is 30 (Urinary problems have a huge specific impact on QoL).
Changes in Female Sexual Function Index (FSFI) and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  The FSFI ("Female Sexual Function Index") is based on questions concerning female sexual functions. It consists of 19 items covering 6 domains, namely sexual desire, arousal (both subjective and physiologic), lubrication, orgasm, satisfaction, and pain. The lowest possible score in the total FSFI is 2 (asymptomatic); the highest possible score is 36 (symptomatic).
Changes in International Index of Erectile Function (IIEF) and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  The IIEF ("International Index of Erectile Function") is based on questions concerning erectile dysfunction. It consists of 15 items covering 5 domains, namely erectile functioning, orgasmic functioning, sexual desire, and intercourse satisfaction along with a fifth component which encompasses the concept of overall sexual satisfaction. While items 1-10 are rated on a 6-point Likert-type scale from 0 to 5, items 11-15 are rated on a 5-point Likert-type scale from 1 to 5. Higher scores are reflecting less dysfunction. Domain scores are computed by summing the sores for individual items in each domain.
Changes in International Spinal Cord Society (ISCoS) Female / Male sexual function data sets and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
Changes in Neurogenic Bowel Dysfunction (NBD) score and their relation to clinical outcomes | Baseline; once per week during the TTNS intervention period; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  The NBD ("Neurogenic Bowel Dysfunction") score is based on questions concerning constipation and fecal incontinence and was developed for and validated in the spinal cord injury population. It consists of 10 items. The lowest possible score in the total NBD is 0 (asymptomatic); the highest possible score is 47 (symptomatic). The interpretation of the total NBD score is very minor NBD (0-6), minor NBD (7-9), moderate NBD (10-13), and severe NBD (≥14).The NBD score is assessed by using the international spinal cord injury (ISCoS) bowel function basic data set.
Volumetric changes during rectal sensitivity testing and barostat assessment and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  Initial sensation [mL], volume at urge to defecate [mL], maximum tolerated volume [mL] as assessed by rectal sensitivity testing; rectal capacity [mL] assessed by barostat assessment
Pressure changes during anorectal manometry and barostat assessment and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  Basal internal anal sphincter pressure [mmHg], squeeze external anal sphincter pressure [mmHg], relaxation internal anal sphincter pressure during defecation [%, mmHg], intraabdominal pressure during defecation [mmHg]
Changes in rectal compliance [mL/cmH2O] during anorectal manometry and barostat assessment and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
Changes in defecatory disorder [Rao's classification] identified during anorectal manometry and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  Anorectal manometry is the preferable test for defecatory disorder. Rao's classification describes the four types of manometric patterns (I-IV) that are identified through manometric assessments
Changes International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) protocol | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) assessment to quantify the severity of the spinal cord injury
Changes in Lower Extremities Motor Scale (LEMS) from International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) protocol | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  LEMS is based on assessments of ISNCSCI and composed from the sum of muscle function grading of the five key muscles of the lower limbs. It consists of a 6-point scale (0=no; 5=normal activity) for each muscle and body site. The lowest possible score in the total LEMS score for one body site is 0 (symptomatic); the highest possible score is 50 (asymptomatic).
Changes in Upper Extremities Motor Scale (UEMS) from International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) protocol | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  UEMS is based on assessments of ISNCSCI and composed from the sum of muscle function grading of the five key muscles of the upper limbs. It consists of a 6-point scale (0=no; 5=normal activity) for each muscle and body site. The lowest possible score in the total LEMS score for one body site is 0 (symptomatic); the highest possible score is 50 (asymptomatic).
Changes in Spinal Cord Independence Measure III (SCIM-III) and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  The SCIM-III ("Spinal Cord Independence Measure III") score is based on questions concerning independence of persons with a spinal cord injured. It consists of 19 items covering 3 domains, self-care, respiration and sphincter management, and mobility. The self-care subscale ranges from 0 to 20. The respiration and sphincter management subscale ranges from 0 to 40. The mobility subscale ranges from 0 to 40. Total score ranges from 0 (symptomatic) to 100 (asymptomatic). Higher scores reflect higher levels of independence.
Changes in spasticity in the knee and elbow flexors and extensors from the Modified Ashworth Scale (MAS) assessment and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  The MAS is a 5-point nominal scale that uses subjective clinical assessments of muscle tone ranging from 0 - 'No increases in tone' to 4 - 'Limb rigid in flexion or extension'. A grade of (1+) indicates resistance in the movement.
Changes in spasticity in daily life as assessed by the Spinal Cord Injury Spasticity Evaluation Tool (SCI-SET) questionnaire and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  The SCI-SET ("Spinal Cord Injury Spasticity Evaluation Tool ") score is based on questions concerning the positive and negative effects of spasticity on different areas of daily life. Each of the 35 items are rated on a 7-point scale (-3=extremely problematic; 0=no effect; 3=extremely helpful). Calculations include counts and sum scores of areas of daily life where spasticity is problematic (count range: 0 to 35, sum score range: 35 to 0) or helpful (counts range: 0 to 35, sum score range: 0 to +35) as well as a mean score of all applicable items (range: -3 to +3)
Changes in neurophysiology measurements of evoked potentials (EPs) as well as nerve conduction measurements and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
Changes in lower urinary tract (LUT) neurophysiology: Current perception thresholds (CPTs) and LUT sensory evoked potentials (LUTSEPs) with their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
Changes in frequency power of surface electromyography (EMG) and electroencephalography (EEG) and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  Fast Fourier Transformation analysis for delta, theta, alpha, beta, and gamma band power as assessed via EEG of the cortex and EMG of the muscle
Changes in EMG and EEG coherence measures and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  Coherence for EEG and EMG signals computed as cortico-muscular, inter- and intra-muscular coherence for typical EEG/EMG frequency bands (delta, theta, alpha, beta, and gamma).
Changes in white and gray matter area in the lumbosacral enlargement (LSE) and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  White and gray matter areas are obtained by segmenting the T2*-weighted MRI images for white and gray matter at the level of LSE
Changes in white and gray matter area in upper cervical cord (at C2/C3) and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  Obtained by segmenting the T2*-weighted MRI images for white and gray matter at the vertebral level C2/C3.
Changes in white and gray matter volume of the conus medullaris (CM) and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  White and gray matter volume are obtained by segmenting the T2*-weighted MRI images for white and gray matter in the CM
Changes in gray and white matter volume in the brain and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  Gray and white matter volume in the brain are computed by feeding the whole-brain T1-weighted MRI images into a voxel-based morphometry algorithm. Changes in the gray and white matter volume will be evaluated in urologically relevant brain areas.
Changes in fractional anisotropy (FA) in the brain and spinal cord and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  FA is a common dimensionless measure used in Diffusion Tensor Imaging (DTI) studies and ranges from 0, isotropic movement of water molecules (e.g., cerebrospinal fluid), to 1, fully anisotropic movement of water molecules (e.g., fiber bundles).
Changes in diffusivity in the brain and spinal cord and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  Mean, axial, and radial diffusivity (MD, AD, RD) are common measures used in DTI studies providing information about the integrity of the underlying tissue.
Changes in brain and spinal cord tissue microstructure and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  Quantitative tissue parameters assessed using MRI Multi-Parameter Mapping.
Expression profile of microRNA (miRNA) in urine and blood as well as their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  MicroRNA (miRNA) sequencing is used to identify regulated miRNAs specific to TTNS intervention in urine and blood.
Changes in inflammatory markers in bladder tissue, blood, and urine, as well as their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
Changes in levels of neurotransmitters (neurotrophins) in blood, and urine, as well as their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  Analysis will be performed using ELISA to detect molecules likely to be involved in the underlying molecular mechanisms of neuromodulation.
Changes in the composition of urinary and stool microbiome and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end
  Gut and bladder microbial patterns are determined from stool and urine samples
Changes in bladder tissue and their relation to clinical outcomes | Baseline; 3 months after SCI; 6 months after SCI; 12 months after SCI / study end

OTHER OUTCOMES:
Incidence of side effects as well as number and intensity/severity (mild/moderate/severe) of adverse events (AEs) and serious adverse events (SAEs) for the following categories: | During complete study period, up to 12 months
  * infection - Urinary Tract Infection (UTI)
  * infection - other than UTI
  * skin irritation at the electrode site
  * irritation-related symptoms (e.g. dysuria, hematuria) immediately following a LUT intervention
  * neuro-urological deterioration
  * pressure ulcer
  * neurological deterioration
  * increase in pain
  * increase in spasticity
  * deep vein thrombosis / pulmonary embolism
  * autonomic dysreflexia
  * transfer/admittance to an acute care facility

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M. Kessler, Prof. Dr. med., Study Chair — University of Zurich; Thomas M. Kessler, Prof. Dr. med., Principal Investigator — Balgrist University Hospital; Armin Curt, Prof. Dr. med., Principal Investigator — Balgrist University Hospital; Martin Brinkhof, Dr., Principal Investigator — Swiss Paraplegic Research, Nottwil; Jürgen Pannek, Prof. Dr. med., Principal Investigator — Swiss Paraplegic Centre
Locations (4):
- Switzerland (4):
  - Department of Neuro-Urology, Spinal Cord Injury Centre & Research, Balgrist University Hospital, Zurich, Canton of Zurich
  - REHAB Basel, Basel
  - Swiss Paraplegic Centre, Nottwil
  - Spinal Cord Injury Department, Clinique romande de réadaption, Sion

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) and data dictionaries that underlie results in a publication are to be uploaded to a public data registry in cases where this can be done without compromising patient privacy. Given the small size of the dataset and that spinal cord injury (SCI) is a rare condition, to ensure identity protection any publicly available dataset(s) will be modified to reduce the number of indirect identifier variables, e.g. continuous variables such as age will be grouped, categorical or binary variables with small group numbers such as study centre will not be provided. When data sets cannot be sufficiently de-identified to be made publicly available, they will be made available upon reasonable request. Data judged to be confidential to participants or the participating study centers will not be released, but efforts will be made to provide scientifically meaningful equivalent information.
Supporting Information: Analytic Code
Time Frame: Post-publication data packages, containing the analysis data set presented in scientific reports will be available starting 6 months after the publication date. Data that are not being prepared for publication will be available to secondary users starting 4 years after study completion or discontinuation. All data will be kept for at least 10 years after study completion or discontinuation.
Access Criteria: Requests for data access will be reviewed by the TASCI steering committee, which includes the four project PIs and representatives from each of the participating study centers. The steering committee will request a project plan, including at a minimum an abstract and a list of author names and roles, from the leaders of all projects wishing to use TASCI study data. Project plans will be evaluated on the basis of scientific validity, and also on whether they include adequate measures to protect patient privacy. Secondary users will be asked to sign a data use agreement.

REFERENCES:
- [Background] Birkhauser V, Liechti MD, Anderson CE, Bachmann LM, Baumann S, Baumberger M, Birder LA, Botter SM, Bueler S, Cruz CD, David G, Freund P, Friedl S, Gross O, Hund-Georgiadis M, Husmann K, Jordan X, Koschorke M, Leitner L, Luca E, Mehnert U, Mohr S, Mohammadzada F, Monastyrskaya K, Pfender N, Pohl D, Sadri H, Sartori AM, Schubert M, Sprengel K, Stalder SA, Stoyanov J, Stress C, Tatu A, Tawadros C, van der Lely S, Wollner J, Zubler V, Curt A, Pannek J, Brinkhof MWG, Kessler TM. TASCI-transcutaneous tibial nerve stimulation in patients with acute spinal cord injury to prevent neurogenic detrusor overactivity: protocol for a nationwide, randomised, sham-controlled, double-blind clinical trial. BMJ Open. 2020 Aug 13;10(8):e039164. doi: 10.1136/bmjopen-2020-039164. PMID 32792454
- [Background] Liechti MD, van der Lely S, Stalder SA, Anderson CE, Birkhauser V, Bachmann LM, Brinkhof MWG, Curt A, Jordan X, Leitner L, Mehnert U, Mohr S, Pannek J, Schubert M, Kessler TM; TASCI Study Group. Update from TASCI, a Nationwide, Randomized, Sham-controlled, Double-blind Clinical Trial on Transcutaneous Tibial Nerve Stimulation in Patients with Acute Spinal Cord Injury to Prevent Neurogenic Detrusor Overactivity. Eur Urol Focus. 2020 Sep 15;6(5):877-879. doi: 10.1016/j.euf.2019.09.019. Epub 2019 Oct 8. PMID 31601539
- [Background] Anderson CE, Birkhauser V, Stalder SA, Bachmann LM, Curt A, Jordan X, Leitner L, Liechti MD, Mehnert U, Mohr S, Pannek J, Schubert M, van der Lely S, Kessler TM, Brinkhof MWG. Optimizing clinical trial design using prospective cohort study data: a case study in neuro-urology. Spinal Cord. 2021 Sep;59(9):1003-1012. doi: 10.1038/s41393-020-00588-z. Epub 2020 Nov 24. PMID 33235299
- [Background] Bueler S, Yiannakas MC, Damjanovski Z, Freund P, Liechti MD, David G. Optimized multi-echo gradient-echo magnetic resonance imaging for gray and white matter segmentation in the lumbosacral cord at 3 T. Sci Rep. 2022 Oct 3;12(1):16498. doi: 10.1038/s41598-022-20395-1. PMID 36192560
- [Background] Bueler S, Freund P, Kessler TM, Liechti MD, David G. Improved inter-subject alignment of the lumbosacral cord for group-level in vivo gray and white matter assessments: A scan-rescan MRI study at 3T. PLoS One. 2024 Apr 16;19(4):e0301449. doi: 10.1371/journal.pone.0301449. eCollection 2024. PMID 38626171
- [Background] Stalder SA, van der Lely S, Anderson CE, Birkhauser V, Curt A, Gross O, Leitner L, Mehnert U, Schubert M, Tornic J, Kessler TM, Liechti MD. Development of a Sham Protocol to Investigate Transcutaneous Tibial Nerve Stimulation in Randomised, Sham-Controlled, Double-Blind Clinical Trials. Biomedicines. 2023 Jul 7;11(7):1931. doi: 10.3390/biomedicines11071931. PMID 37509569
- [Background] Beghini L, Bueler S, Liechti MD, Jaffray A, David G, Vannesjo SJ. Optimized navigator-based correction of breathing-induced B0 field fluctuations in multi-echo gradient-echo imaging of the spinal cord. Magn Reson Med. 2025 Jul;94(1):215-230. doi: 10.1002/mrm.30475. Epub 2025 Mar 4. PMID 40034000
- [Background] Bueler S, Anderson CE, Birkhauser V, Freund P, Gross O, Kessler TM, Kundig CW, Leitner L, Mahnoor N, Mehnert U, Rothlisberger R, Stalder SA, van der Lely S, Zipser CM, David G, Liechti MD. Remote neurodegeneration in the lumbosacral cord one month after spinal cord injury: a cross-sectional MRI study. Ann Clin Transl Neurol. 2025 Mar;12(3):523-537. doi: 10.1002/acn3.52298. Epub 2025 Jan 27. PMID 39869509
- See also: TASCI on Swiss National Science Foundation grant database — http://p3.snf.ch/project-179644